CLINICAL TRIAL: NCT02006602
Title: An Open-label, Randomised, Single Dose, Two-way Crossover Pilot Study to Determine the Relative Bioavailability of One 16mg Tablet Formulation of Candesartan Cilexetil (GW615775) Relative to One 16mg Reference Tablet of Candesartan Cilexetil (Atacand) in Healthy Adult Human Subjects Under Fasting Conditions
Brief Title: Bioavailability Study of Candesartan Cilexetil 16mg Tablet Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201011
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Hypertension
Keywords: Candesartan cilexetil; Healthy adult human subjects; Bioequivalence
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 reference then test (Experimental): Subjects will be randomized and receive the following two treatments administered orally in a fasting state: A=Single dose of candesartan cilexetil (Reference treatment) 16mg; B= Single dose of candesartan cilexetil (Test formulation) 16mg. The two treatment periods will be separated by a washout period of at least 7 days and no more than 14 days.
  Interventions: Drug: Candesartan cilexetil (GW615775, Test formulation); Drug: Candesartan cilexetil (Reference treatment)
- Arm 2 test then reference (Experimental): Subjects will receive the following two treatments administered orally in a fasting state: A= Single dose of candesartan cilexetil (Test formulation) 16mg. B=Single dose of candesartan cilexetil (Reference treatment) 16mg. The two treatment periods will be separated by a washout period of at least 7 days and no more than 14 days.
  Interventions: Drug: Candesartan cilexetil (GW615775, Test formulation); Drug: Candesartan cilexetil (Reference treatment)

INTERVENTIONS:
Drug: Candesartan cilexetil (GW615775, Test formulation) — Test formulation candesartan cilexetil 16 mg will be supplied as round, biconvex white tablets with PX 16 embossed in one face and scored in the other face.
Drug: Candesartan cilexetil (Reference treatment) — Reference treatment of candesartan cilexetil 16 mg will be supplied as round, biconvex pink tablets, scored in one face and with embossment in both faces (016 embossment in the plain face and A CH in the scored face).

SUMMARY:
This will be an open-label, randomized, single dose, two-way crossover study. Each subject will participate in both treatment periods and will receive single oral doses of candesartan cilexetil (GW615775) and reference candesartan cilexetil (ATACAND™); the treatment periods will be separated by a washout period of at least 7 days and no greater than 14 days. This study aims to determine the relative bioavailability of a 16mg test formulation tablet of candesartan cilexetil (GW615775) compared to an 16mg reference tablet of candesartan cilexetil in healthy adult subjects. ATACAND is a registered trademark of the Astra/Zeneca group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Male and females aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the GSK Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 50kg and body mass index within the range 19 - 24.9 kilogram per square meter (kg/m^2) (inclusive).
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records; or postmenopausal defined as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli-international units (MIU) per milliliter (mL) and estradiol <40 pigogram per mL (pg/mL) (<147 picomole per liter) is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method; Child-bearing potential with negative pregnancy test as determined by serum and urine human chorionic gonadotropin (hCG) test at screening or prior to dosing and Agrees to use one of the contraception methods listed in Protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up contact visitor has only same-sex partners, when this is her preferred and usual lifestyle.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Protocol. This criterion must be followed from the time of the first dose of study medication until the follow-up contact visit.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Alanine transaminase, alkaline phosphatase and bilirubin <= 1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on single or averaged corrected QT interval (QTc) of triplicate electrocardiograms (ECGs) obtained over a brief recording period: QT duration corrected for heart rate by Fridericia's formula (QTcF) <450 milliseconds (msec).

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Gastrointestinal disease or with gastrointestinal surgical history which can affect the absorption of the investigational drug.
* Any subject with a systolic blood pressure (BP) <95 millimeters of mercury (mmHg) or with a recent history of postural symptoms
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive pre-study drug/alcohol screen.
* A positive test for Human immunodeficiency virus (HIV) antibody.
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-12-13 (Actual); Primary Completion 2014-01-22 (Actual); Study Completion 2014-01-22 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic (PK) parameters assessed by Cmax, AUC(0-infinity) and AUC(0-t) | Pre-dose, 0.5 hour (hr), 1 hr, 1.5 hr, 2 hr, 2.5 hr, 3 hr, 3.5 hr, 4 hr, 4.5 hr, 5 hr, 5.5 hr, 6 hr, 7 hr, 8 hr, 10 hr, 12 hr, 16 hr, 24 hr, 36 hr and 48 hr of each treatment period.
  PK parameters include: Maximum observed concentration (Cmax), area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0 infinity]) and area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments [AUC(0 t)].

SECONDARY OUTCOMES:
PK parameters assessed by tmax, %AUCex and t1/2 | Pre dose, 0.5 hr, 1 hr, 1.5 hr, 2 hr, 2.5 hr, 3 hr, 3.5 hr, 4 hr, 4.5 hr, 5 hr, 5.5 hr, 6 hr, 7 hr, 8 hr, 10 hr, 12 hr, 16 hr, 24 hr, 36 hr and 48 hr of each treatment period.
  PK parameters include: Percentage of AUC(0-infinity) obtained by extrapolation (%AUCex), time of occurrence of Cmax (tmax), terminal phase half-life (t1/2).
Safety and tolerability assessment as assessed by adverse events (AEs) | Up to 35 days
Safety and tolerability assessment as assessed by vital signs | Up to 35 days
  Vital sign measurements will include systolic and diastolic blood pressure, and pulse rate.
Safety and tolerability assessment as assessed by clinical laboratory values | Up to 35 days
  Clinical laboratory assessments will include hematology, clinical chemistry, routine urinalysis and additional parameters.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hyderabad, India

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 201011 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/201011?search=study&search_terms=201011#rs
- Available data/document: Informed Consent Form: 201011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 201011 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register